CLINICAL TRIAL: NCT06590662
Title: A Randomized, Double-blind, Placebo-controlled Trial Comparing the Efficacy and Tolerance of Solriamfetol in Patients Affected with Idiopathic Hypersomnia.
Brief Title: Efficacy and Tolerance of Solriamfetol in Patients Affected with Idiopathic Hypersomnia.
Acronym: SOLR-IH
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RECHMPL23_0432
Record Dates: First submitted 2024-08-06; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Idiopathic Hypersomnia
Keywords: Idiopathic hypersomnia; Solriamfetol; polysomnography
MeSH Terms: conditions — Idiopathic Hypersomnia | interventions — solriamfetol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Solriamfetol (Experimental): Solriamfetol will be taken once a day upon awakening during 7-weeks
  Interventions: Drug: Solriamfetol
- Placebo (Placebo Comparator): Placebo will be taken once a day upon awakening during 7-weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Solriamfetol — Patient with a diagnostic of idiopathic hypersomnia (ICSD-3 criteria) will be randomized to receive solriamfetol or placebo for 7 weeks of treatment period. For the experimental arm, the dose will be progressively increased beginning at 75 mg to 300 mg according to tolerance to treatment.
  Solriamfetol will be taken once a day upon awakening Schema of dispensation
  1. One tablet of solriamfetol 75 mg per day for 1 week (week 1)
  2. 150 mg of solriamfetol per day for 2 weeks (weeks 2 and 3)
  3. According clinical judgment, Dose either maintained stable at 150 mg or increased to 300 mg per day for 2 weeks (weeks 4 and 5).
  4. Prescription at week 5: Dose maintained at 150 or 300 mg or reduced at 150 mg per day according to benefit and safety for 2 weeks.
  Treatment duration: 7 weeks treatment period.
  Arms: Solriamfetol
Drug: Placebo — Patient with a diagnostic of idiopathic hypersomnia (ICSD-3 criteria) will be randomized to receive solriamfetol or placebo for 7 weeks of treatment period.
  Placebo will be taken once a day upon awakening Schema of dispensation
  1. One tablet of placebo per day for 1 week (week 1)
  2. Two tablets of placebo per day for 2 weeks (weeks 2 and 3)
  3. According clinical judgment, Either maintained stable with 2 tablets or increased to 4 tablets per day for 2 weeks (weeks 4 and 5).
  4. Prescription at week 5: Dose maintained at 2 or 4 tablets or reduced at 2 tablets per day according to benefit and safety for 2 weeks.
  Treatment duration: 7 weeks placebo period.
  Arms: Placebo

SUMMARY:
This Phase II clinical trial is a monocenter, double-blind, randomized, placebo-controlled study aimed at evaluate the efficacy and safety of solriamfetol from 75 to 300 mg per day in IH patients.

Patients will be randomized (1:1) to receive either solriamfetol or placebo, with titration, every morning upon awakening during all treatment periods (Day 0 to Week 7).

ELIGIBILITY:
Main inclusion criteria:

* Age between 18 and 60 years-old
* BMI between 18 and 30 kg/m2
* Diagnostic of idiopathic hypersomnia (ICSD-3 criteria) made in the last 5 years, based on Polysomnography (PSG) and Multiple Sleep Latency Test (MSLT) results, showing either: a mean sleep latency (MSL) of ≤8 minutes and < 2 SOREMPs and/or a 24-h long term polysomnography recording showing total sleep time >11h/24 hours.
* Apnea-hypopnea index (AHI) <15/hour, Apnea index <10/hour, micro-arousals index <15/hour, Periodic limb movement (PLM) index associated with micro-arousals <15/hour on the PSG and MSLT performed within the past 5 years.
* Absence of sleep deprivation, assessed by actigraphy or sleep logs for the 7 days preceding study inclusion
* ESS score ≥11 points
* Written informed consent
* National health insurance coverage
* Understand, read and speaks French well
* The participant agrees to follow the contraceptive requirements detailed in the protocol.

Main non-inclusion criteria

* Non-stabilized hypertension
* To be at imminent risk of suicide or injury to self, others, or property, or the participant has attempted suicide within the past year before screening, or has positive answers on items number 4 or 5 on the Colombia-Suicide Severity Rating Scale (based on the 6 months before randomization).
* Other psychiatric conditions in the past 6 months
* Presence of other central nervous system diseases: neurodegenerative diseases, seizure disorders, or history of head trauma associated with loss of consciousness
* Prior history of psychotic episodes
* Psychostimulant treatment with modafinil, methylphenidate, mazindol, pitolisant, ongoing or within 15 days prior to visit 1
* Treatment for obstructive sleep apnea-hypopnea syndrome ongoing or within 15 days prior to visit 1
* Treatment with psychotropic drugs: neuroleptics (i.e. clozapine, olanzapine, aripiprazole, …), sedative hypnotics (benzodiazepines, zolpidem, zopiclone), central nervous system depressants (barbiturates, …), antidepressants (SSRI (e.g. fluoxetine, sertraline, paroxetine…), serotonin and norepinephrine reuptake inhibitors (SRNI : e.g. venlafaxine, duloxetine), Monoamine oxidase inhibitors), anxiolytic drugs, anticonvulsive therapy (i.e. topiramate, inhibitors of GHB dehydrogenase (i.e. valproate, ethosuximide, phenytoin), or drugs for pain (level 2 (e.g. codeine, tramadol), and level 3 (morphine and derivatives)), ongoing or within 30 days prior to visit 1.
* Treatment with dopamine antagonist antiemetics except domperidone, Catechol-O-methyltransferase (COMT) inhibitors, or sedative antihistamines ongoing or within 30 days prior to visit 1

  => Of note, for all the above treatments: if patient has received such therapy, a washout-period of at least 15 days, or equivalent to 5 half-lives of the drug, prior to the inclusion in the study is required before starting treatment in this study. Of note, for antidepressants, a washout of at least 30 days should be required.
* Previously treated with solriamfetol
* History of chronic alcohol or drug abuse within the prior 12 months
* Malignant neoplastic disease requiring therapy within 12 months prior to Visit 1 or clinically relevant
* Heart failure, unstable hypertension or other cardiovascular disease compromising the patient's wellbeing or ability to participate in this study
* Renal or hepatic impairment
* No regular sleep at night: shift work or other continuous non-disease-related life conditions
* Has received any other investigational drug within 30 days or 5 half-lives (whichever is longer) prior to screening or plans to use an investigational drug (other than the study intervention) during the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2026-11-15 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Idiopathic hypersomnia severity scale (IHSS) score | From baseline to week 7
  IHSS is a tool used to measure the severity of the symptoms experienced by patients with IH during the previous month. The IHSS includes 2 items (1 and 2) on nighttime sleep duration and quality, 3 items (3, 4, and 5) on sleep inertia and sleep drunkenness after nighttime sleep and 1 (8) after daytime nap, and 3 items (6, 7, and 9) on diurnal symptoms (nap occurrence, daytime sleepiness). Items 10-14 assess daytime functioning alterations due to hypersomnolence. Six items are scored on a 3-point Likert scale and 8 items on a 4-point Likert scale; the Likert scale is a point scale that is used to allow the individual to express how much they agree or disagree with a particular statement. The total IHSS score is the sum of all item scores (range: 0-50), and higher scores indicate more severe symptoms.

SECONDARY OUTCOMES:
Epworth Sleepiness Scale (ESS) score | From baseline to week 7
  ESS is a short 8-item questionnaire designed to assess daytime sleepiness. Participants assign a score from 0 to 3 (0 = never; 1 = weak; 2 = moderate; 3 = strong).The minimum score is 0 and the maximum score is 24.
Maintenance of Wakefulness Test (MWT) | From baseline to week 7
  MWT is used in this study to assess an individual's ability to maintain awake while resisting the pressure to fall asleep. Patients will be administrated four 40-minute MWT session at 2 hours interval at baseline visit 2 (Day 14) and at endpoint visit (Day 35), according to validated standard. The changes in MWT will be compared between the treatment groups.
Psychomotor vigilance task (PVT) | From baseline to week 7
  PVT is a widely utilized as a measure of behavioral alertness, primary due to its high sensitivity to sleep deprivation and its psychometric advantages over other cognitive tests. The standard 10-min PVT measures sustained or vigilant attention by recording response times (RT) to visual (or auditory) stimuli presented at random inter-stimulus intervals.
Karolinska Sleepiness Scale (KSS) | From baseline to week 7
  KSS measures the subjective level of sleepiness at a particular time during the day. On this scale subjects indicate which level best reflects the psycho-physical sate experienced in the last 10 min. The KSS is a measure of situational sleepiness.
Sleep inertia questionnaire | From baseline to week 7
  The Sleep inertia questionnaire evaluated self-reported sleep inertia and sleep drunkenness on the day of the PVT assessment, utilizing wording similar to items from IHSS scale to assess their presence and duration.
Clinical Global Impression Scale for Change (CGI-C) | From baseline to week 7
  CGI-C was used to measure, the change in excessive daytime sleepiness (EDS) compared to baseline. This scale if administrated by the same investigator and consists of a 7-grade scale as follows: "very much improved", "much improved", "minimally improved", "no change", "minimally worse," "much worse", "very much worse".
Clinical Global Impression Scale for Severity (CGI-S) | From baseline to week 7
  CGI-S is an observer-rated scale that measures illness severity by using a 7- grade scale ranging from ("normal, not at all ill") "borderline ill", "slightly ill", "moderately ill", "markedly ill", "severely ill", "among the most extremely ill patients".
The EuroQol 5-Dimensional Descriptive System (EQ-5D-3L) | From baseline to week 7
  EQ-5D-3L is a validated generic quality of life questionnaire that can be completed by the patient and/or caregiver and assesses 5 dimensions: mobility, washing and dressing, daily living activities, discomfort/pain, and anxiety. Each question has 3 response levels: no problem, some problems and important problems. The questionnaire includes also a visual analog scale in which the patient quantifies his or her perception of quality of life using a score ranging from the worst imaginable state of health (0) to the best imaginable state of health (100).
Work Productivity and Activity Impairment- General Health (WPAI:GH) | From baseline to week 7
  WPAI:GH is a well validated instrument to measure the effect of health conditions on work productivity and daily activities. The WPAI-GH consists of six questions: 1 = currently employed; 2 = hours missed due to health problems; 3 = hours missed other reasons; 4 = hours actually worked; 5 = degree health affected productivity while working (using a 0 to 10 Visual Analogue Scale (VAS)); 6 = degree health affected productivity in regular unpaid activities (VAS).
Questionnaire on Functional Outcomes of Sleep | From baseline to week 7
  FOSQ consists of 10 questions related to the effects of fatigue on daily activities. Each item in the FOSQ is rated on a 4 to 6-point scale, where patients provide their level of agreement of frequency of occurrence specific statements to their functioning.
Logbook for compliance to monitor | From baseline to week 7
  The patient logbook must be completed throughout the treatment to monitor compliance with treatment.
Percentage of sleep stages | From baseline to week 7
  % of time spent in stage 1 and 2 sleep stages and stage 3 during polysomnography
Microarousal index | From baseline to 7 weeks
  Microarousal index is apneas + hypopneas per hour of sleep during polysomnography assessment. When the respiratory event index (apneas + hypopneas per hour of sleep) is between 5 and 15 per hour of sleep, SAS is considered mild, and between 15 and 30, moderate. Above 30, it is severe.
Total sleep time | From baseline to 7 weeks
  Total sleep time measured in minutes during polysomnography

OTHER OUTCOMES:
24-hour Ambulatory Blood Pressure Monitoring (ABPM) | From baseline to week 8
  24-hour ABPM is an accurate, fully automated, and non-invasive method for evaluation of the 24-hour hemodynamic profile of a subject by multiple and regular blood pressure and heart rate measurements. The ABPM will be monitored at baseline and just before the end visit.
Actigraphy to detect the wake and sleep cycle | From 1 week before baseline to 1 week before week 7
  Actigraphy is a non-invasive test carried out using a device worn on the wrist over a period of one week. It aims to detect the pattern of waking and sleeping.
Pregnancy test (beta HCG blood test) | 90 days before baseline
  The dosage taken during a pregnancy test is the beta-HCG dosage. This dosage is carried out from a blood test. It is not necessary to be fasting to take the exam.

CONTACTS AND LOCATIONS:
Overall Officials: Yves DAUVILLIERS, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University Hospital of Montpellier, Montpellier, France